CLINICAL TRIAL: NCT01318746
Title: The Circadian Rhythm of Potassium and Cystatin c and the Day-to-day Variability
Brief Title: The Circadian Rhythm of Potassium and Cystatin C
Acronym: Potassium
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 4408
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Cardiac Arrhythmias; Sudden Cardiac Death
Keywords: change of potassium amount, circadian and day-to-day variability
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy group: 15 persons with normal renal function
  Interventions: Procedure: Blood withdrawal
- Renal failure: 15 persons with renal failure (GFR < 60 ml/min)
  Interventions: Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Blood withdrawal — blood withdrawal every 2 hours during 24 hours

SUMMARY:
The potassium value is important to prevent cardiac arrhythmias and sudden cardiac death. In patients with renal failure, the potassium value is not stable and tends to raise. Until now there are no data available if the potassium value has a circadian rhythm and if there are individual changes from day to day.

DETAILED DESCRIPTION:
Potassium and cystatin c is measured every 2 hours during 24 hours, twice. There are two groups of patients: Patients with eGFR < 60 ml/min and patients with eGFR > 60 ml/min

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* normal renal function and impaired renal function (GFR < 60 ml/min) respectively

Exclusion Criteria:

* pregnancy
* anaemia (Hb<10 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy persons compared to patients with renal failure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Potassium rhythm | twice in 24 hours
  15 persons with normal renal function are hospitalized for 24 hours. Blood samples are taken every 2 hours in order to investigate the potassium value.
  It is repeated with 5 persons after 2 days, with 5 persons after 4 and with 5 persons after 6 days.

SECONDARY OUTCOMES:
Potassium value in renal failure | twice in 24 hours
  15 persons with renal failure (GFR < 60 ml/min) are hospitalized for 24 hours. Blood samples are taken every 2 hours in order to investigate the potassium value It is repeated with 5 persons after 2 days, with 5 persons after 4 and with 5 persons after 6 days.

CONTACTS AND LOCATIONS:
Overall Officials: Roland E. Schmieder, MD, Principal Investigator — Department of Nephrology and Hypertension, University of Erlangen-Nürnberg Medical School
Locations (1):
- Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen, Germany

REFERENCES:
- [Result] Schmidt ST, Ditting T, Deutsch B, Schutte R, Friedrich S, Kistner I, Ott C, Raff U, Veelken R, Schmieder RE. Circadian rhythm and day to day variability of serum potassium concentration: a pilot study. J Nephrol. 2015 Apr;28(2):165-72. doi: 10.1007/s40620-014-0115-7. Epub 2014 Jul 3. PMID 24990164